CLINICAL TRIAL: NCT07286851
Title: Effects of Topical Neomycin on Skin Graft Outcomes in Rural Bangladesh: a Retrospective Cohort Study
Brief Title: Do Topical Antibiotics Improve Skin Graft Results?
Status: Completed | Type: Observational
Sponsor: LAMB Project (Other)
Responsible Party: Principal Investigator, Jonathan Egle, General Surgeon, Deputy Medical Director, LAMB Project
Other Study IDs: REC2025/03
Record Dates: First submitted 2025-12-02; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Skin Transplantation; Wounds and Injuries; Antibiotic Prophylaxis Surgery
Keywords: bangladesh; developing countries
MeSH Terms: conditions — Wounds and Injuries | interventions — Neomycin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Patients who had skin graft procedure before the topical antibiotic protocol was initiated
- Neomycin: Patients who had skin graft procedure after the topical antibiotic protocol was initiated. Patients had topical neomycin applied at the time of their surgeries.
  Interventions: Drug: Neomycin

INTERVENTIONS:
Drug: Neomycin — Topical neomycin was applied at the time of split-thickness skin graft surgery.
  Groups: Neomycin

SUMMARY:
The goal of this study is to see if putting antibiotic ointment on a skin graft when the surgery is being done helps prevent the skin graft from getting infected after the operation. The study is looking at all skin grafts done in a rural Bangladesh hospital.

The main questions it aims to answer are:

Does the antibiotic lower the number of infections that happen? Does the antibiotic make the overall outcome of the skin graft better? Do patients who get the antibiotic need fewer extra surgeries?

Researchers will compare the outcomes from patients who had skin grafts before the hospital started applying antibiotic ointment to the outcomes of patients after the hospital began applying antibiotic ointment.

Participants who have already had their skin graft treatment completed will have their medical records reviewed by researchers. The outcomes of their treatment will be written down.

ELIGIBILITY:
Inclusion Criteria:

* patient undergoing a split-thickness skin graft at the hospital where research is conducted

Exclusion Criteria:

* Missing or incomplete medical record

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with wounds undergoing split-thickness skin graft surgery at a single rural hospital in Bangladesh.
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Post-operative infection rate | Measured if present at any time during the patient's initial post-operative hospitalization, which averaged 20 days, from time of operation until time of discharge.
  Whether patients had post-operative infection during their hospitalization, classified as "yes" or "no" as defined by any of the following being present: "post-operative infection" diagnosis written in the patient's medical record, change or increase in antibiotic therapy post-operatively, or the presence of pus documented at the skin graft site.

SECONDARY OUTCOMES:
Skin graft take | Measured at the time of discharge from the patient's initial post-operative hospitalization, which averaged 20 days.
  Percentage of skin graft that remained intact at the time of discharge, as estimated by the treating surgeon and documented in the patient's record.
Need for operative re-intervention | From the time of operation until the end of the study period (up to three years for the earliest skin graft patients).
  Whether patient needed to return to the operating room for additional procedures (such as debridement or repeat skin grafting) for the same wound, classified as "yes" or "no."
Length of stay | Measured at the time of discharge from the patient's initial post-operative hospitalization, which averaged 20 days.
  Number of days spent in the hospital during the initial post-operative period.
Allergic reaction | Measured if present at any time during the patient's initial post-operative hospitalization, which averaged 20 days, from time of operation until time of discharge.
  Whether patient had any allergic reaction to neomycin or any other substance documented - categorized as "yes" or "no," based on the new presentation of rash or pruritis.

CONTACTS AND LOCATIONS:
Locations (1):
- LAMB Hospital, Parbatipur, Dinajpur, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication may be available upon reasonable request if the study is published in a peer-reviewed journal.
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: This IPD will be available beginning when the study is published and will be available while the authors continue to be affiliated with the institution where the study has taken place.
Access Criteria: The request for sharing of data must be reviewed by the LAMB Project Research Ethics Committee, which will make all final decisions about the sharing of individual patient data.